CLINICAL TRIAL: NCT06729034
Title: A Single-center Blinded Crossover Study Investigating the Efficacy of Apixaban in Patients with Painful Venous Malformations with Localized Intravascular Coagulation
Brief Title: A Study of Direct Oral Anticoagulants in Patients with Painful Venous Malformations with Localized Intravascular Coagulation
Acronym: AVA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Nina Haagenrud Schultz, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-511930-11-00; 2024-511930-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-30; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Venous Malformation, Low Flow; Anticoagulants
Keywords: apixaban; venous malformation; localized intravascular coagulation
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Randomized study, crossover design, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study in which participants/care providers/investigators/outcomes assessors are blinded to study intervention.. In case of an emergency, the investigator has the responsibility for determining if unblinding of a participant's intervention assignment is warranted. Participant safety must always be the first consideration in making such a determination. The participant will be carrying a card with contact information of investigator and the medical monitor. The card will be in Norwegian and in English and inform that the person is part of a blinded trial and that he/she may be under anticoagulation with apixaban. In case of major bleeding, the investigator must be contacted who may unblind the participant so that emergency treatment can be considered. In case of a life-threatening bleed, there is no time for contacting the investigator. Then measures must be taken as if the participant is under anticoagulation treatment with apixaban
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban (Experimental): Apixaban 5 mg twice daily
  Interventions: Drug: Apixaban (Eliquis)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban (Eliquis) — 5 mg twice daily
  Arms: Apixaban
Drug: Placebo — placebo twice daily
  Arms: Placebo

SUMMARY:
There are two parts of the study. In Part 1, the invesitgaotrs want to investigate whether treatment with apixaban improves pain and quality of life in patients with painful venous malformations The participants are randomized to different treatment orders of the two treatment periods with apixaban and placebo. Arm 1 starts apixaban followed by placebo and arm 2 starts with placebo followed by apixaban. Between the treatment sequences there will be a washout period of minimum one week.

The participants will register pain and use og pain medication in a diary every day for one week before start of treatment and before evaluation of effect. Also, a quality of life form will be filled out before each consultation.

In Part 2, the investigators will investigate long-term effect and safety of apixaban and reduce dose after 3 months to find the minimal effective dose.

Part 2 includes participants from Part 1 study who experienced effect of treatment or who agree to continue apixaban treatment. Study start of Part 2 is at the end of Part 1. All participants receive the same dose of apixaban as in part 1 (5 mg twice daily), and after 3 months (visit 2) the dose is reduced to 2.5 mg twice daily.

DETAILED DESCRIPTION:
There are no established universal guidelines on the hematologic management of patients with venous malformations (VM) with and without localized intravascular coagulopathy (LIC). Anticoagulation treatment with low molecular weight heparin (LMWH) has improved functionality and decreased pain in patients with VM with localized LIC.

The aim is to study the effect of the direct oral anticoagulant apixaban in patients with painful venous malformations with localized intravascular coagulation.

Apixaban is an oral direct acting anticoagulant shown to be as effective and safe as LMWH and warfarin in treating venous thrombosis.

single-center, prospective double-blind crossover superiority study including patients with venous malformations at age 18-85 years. The participants are randomized to different treatment orders of the two treatment periods with apixaban and placebo. Masking of participants and study personell. Randomization at screening to arm 1 or arm 2. Arm 1 starts apixaban followed by placebo and arm 2 starts with placebo followed by apixaban. Between the treatment sequences there will be a washout period of one week.

Part 2: The AVA Long study is an open-label observational study including participants from the AVA study who experienced effect of treatment or who agree to continue apixaban treatment. Study start of AVA long (part 2) is at study end of part 1. The participants receive the dose of apixaban as in part 1 (5 mg twice daily), but open-label, and after 3 months (visit 2) the dose is reduced to 2.5 mg twice daily. The investigators will investigate long-term efficacy and safety of apixaban and find the minimal effective dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant must be 18-85 years of age at the time of signing the informed consent form (ICF).

  2. Participants who have simple VM with LIC. VM must be diagnosed by MRi and LIC is defined as d-dimer > 2 x upper reference area (21).

  3. Patients must experience pain from the malformation, NRS ≥4. Pain is defined as local pain in the malformation, and the participant must have pain that inhibits daily activity or pain during nighttime that interferes with sleep.

  4. Body weight over 50 kg. 5. Pregnancy test at time of inclusion must be negative 6. Capable of giving written informed consent

Exclusion Criteria:

1. History of major bleeding, known disease of the GI tractus with risk of bleeding (ulcera, IBD, tumor), known hemostatic disorder/hemophilia, bariatric surgery or other condition resulting in impaired adsorption of drug, active cancer
2. Lesion or condition if considered a significant risk factor for major bleeding. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities
3. Current treatment with platelet inhibitor, any other anticoagulation treatment e.g. unfractionated heparin, low molecular weight heparin (dalteparin, enoxaparin), heparin derivates (fondaparinux), oral anticoagulants (warfarin, dabigatran, rivaroxaban, edoxaban), NSAIDs, cancer therapy with chemotherapy
4. Current treatment with sirolimus
5. Current treatment with azole-antimycotics (e.g., ketoconazole, itraconazole, voriconazole and posaconazole)
6. Current treatment with HIV protease inhibitors (e.g., ritonavir)
7. Weight <50 kg
8. Known hypersensitivity to the active substance or to any of the excipients listed in the SmPC.
9. Impaired renal function (eGFR < 50 ml/min)
10. Impaired liver function, INR > 1.3 or aminotransferases > 3 times upper limit
11. Pregnancy or breastfeeding
12. Low platelet count (<100 x 109/mL)
13. Any condition that in the view of the investigator would suggest that the patient is unable to comply with the study protocol and procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between apixaban and placebo in change of self-reported pain intensity before and 8 weeks after starting treatment Change in type, dose and frequency of pain medication | From enrollment to the end of treatment at 8 and 17 weeks
  Average numeric rating scale (NRS) score(score 0-10 where 0 represents no pain and 10 represents worst imaginable pain) last 7 days before assessment
Change in pain medication | From enrollment to the end of treatment at 8 and 17 weeks
  Registration of type, dose and frequency of pain medication last 7 days before assessment

SECONDARY OUTCOMES:
Difference between apixaban and placebo in change of quality of life before and 8 weeks after starting treatment | From enrollment until end of treatment, at 8 and 17 weeks
  Outcome Measure for Vascular Malformation (OVAMA) questionnaire
Difference between apixaban and placebo in change of quality of life before and 8 weeks after starting treatment | From enrollment until end of treatment, at 8 and 17 weeks]
  Short form survey-36 (SF-36)
Difference between apixaban and placebo in change in coagulation parameters before and 8 weeks after | From enrollment until after end of treatment at 8 and 17 weeks
  D-dimer
Change in pain intensity after 3 months treatment | From enrollment of Part 2 until completion of treatment at 6 months
  Numeric rating scale (NRS) score at time of evaluation (score 0-10 where 0 represents no pain and 10 represents worst imaginable pain)
Change in pain intensity three months after reducing dose | At changing dose at 3 months after enrollment of Part 2 and after 6 months ( end of treatment)
  Numeric rating scale (NRS) score at time of evaluation (score 0-10 where 0 represents no pain and 10 represents worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data protection regulations does not allow sharing individual participant data

REFERENCES:
- [Background] Liu H, Hu L, Yang X, Xu Z, Gu H, Chen H, Lin X. Dabigatran etexilate is efficacious in consumptive coagulopathy and pain associated with venous malformations. J Vasc Surg Venous Lymphat Disord. 2023 Mar;11(2):397-403.e1. doi: 10.1016/j.jvsv.2022.09.015. Epub 2022 Oct 31. PMID 36328137